CLINICAL TRIAL: NCT00327600
Title: A Phase 1/2 Trial of Amplimexon® (Imexon, Inj.) Plus Dacarbazine (DTIC) in Chemotherapy Naive Patients With Unresectable Stage III or Stage IV Malignant Melanoma
Brief Title: Safety and Efficacy Trial of Imexon Plus DTIC in Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Evan Hersh, VP Medical Affairs, AmpliMed Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-005; NCT00301132 (obsolete NCT alias)
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imexon + DTIC (Experimental)
  Interventions: Drug: imexon; Drug: DTIC

INTERVENTIONS:
Drug: imexon
Drug: DTIC

SUMMARY:
AMP-005 is a Phase 1b/2 clinical trial designed to evaluate whether the new drug, imexon, can be administered in combination with the approved drug, dacarbazine (DTIC), for the treatment of patients with stage III or IV inoperable melanoma. The Phase 1b part of the study is designed to determine whether the two drugs can be safely combined together, and the Phase 2 part of the study is designed to provide additional safety data and to gain an understanding of whether adding imexon to DTIC can improve the outcome for melanoma patients versus the findings from prior clinical studies of DTIC alone.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma; inoperable stage III or IV disease.
* Able to perform the activities of daily living.
* A projected life expectancy of at least 4 months.
* If female, neither pregnant nor nursing.
* Willing to use contraceptives to prevent pregnancy.
* Blood cell counts and blood chemistries in or near normal range.
* Prior radiation is permitted.
* No other serious illnesses.
* No other active malignancy.
* No serious infections.
* No other current drug therapy for the cancer or steroid therapy.

Exclusion Criteria:

* No prior chemotherapy for the stage III or IV disease.
* Brain metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximally tolerated dose of imexon plus DTIC
determine the toxicity and tolerability of the combination
determine response rate and progression free survival

SECONDARY OUTCOMES:
Determine effects of the drug combination on plasma thiol levels and other biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Evan Hersh, MD, Study Director — AmpliMed Corporation
Locations (11):
- United States (11):
  - Investigational Site 009, Los Angeles, California
  - Investigational Site 002, Santa Monica, California
  - University of CO Anschutz Cancer Pavilion, Aurora, Colorado
  - US Oncology Orlando, Cancer Centers of FL, Ocoee, Florida
  - US Oncology Albany, New York Oncology, Albany, New York
  - US Oncology Kettering, Kettering, Ohio
  - US Oncology Greenville, Cancer Centers of the Carolinas, Greenville, South Carolina
  - US Oncology, Tyler Cancer Center, Tyler, Texas
  - Investigational Site 012, Salt Lake City, Utah
  - US Oncology, Virginia Oncology Assoc, Norfolk, Virginia
  - US Oncology Spokane, Cancer Care Northwest, Spokane, Washington

REFERENCES:
- [Result] Weber JS, Samlowski WE, Gonzalez R, Ribas A, Stephenson J, O'Day S, Sato T, Dorr R, Grenier K, Hersh E. A phase 1-2 study of imexon plus dacarbazine in patients with unresectable metastatic melanoma. Cancer. 2010 Aug 1;116(15):3683-91. doi: 10.1002/cncr.25119. PMID 20564083